CLINICAL TRIAL: NCT03541460
Title: Detection of Epigenome Variation Associated With Longevity Among the Multi Ethnic Centenarian Population in Israel
Brief Title: Israeli Multi Ethnic Centenarian Project
Acronym: IMECP
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Israel Science Foundation (Other)
Responsible Party: Principal Investigator, Tzvi Dwolatzky, Director of Geriatric Medicine, Rambam Health Care Campus
Other Study IDs: 0312-14-RMB
Record Dates: First submitted 2017-01-10; First posted 2018-05-30 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: LONGEVITY 1
Keywords: centenarians; epigenome; longevity; healthy aging; epigenetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Three 10 ml blood samples will be drawn into vacutainer tubes (Yellow top with anticoagulant; speckled top without anticoagulant). Blood samples will be analyzed for the levels of hemoglobin, hematocrit, white blood cell counts, and levels of glucose, insulin, albumin, inflammatory markers, and plasma lipids. CD34+Lin- cells will be isolated from the peripheral blood specimen using immuno-magnetic separation technique, followed by cell sorter. Mononuclear cells are separated by Ficoll-Paque density gradient, and CD34+ cells obtained by positive immuno-magnetic bead selection, using Macs columns (Miltenyi Biotech). The purified cells are then subjected to a cell sorter following immunostaining. The isolated cells will be cryopreserved in 10% DMSO by controlled rate freezing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Older Cohort: Demographic, health and functional data will be collected from subjects 95 years and older by means of a structured interview. Blood will be collected for laboratory and genetic testing.
- Younger Controls: Demographic, health and functional data will be collected from the children of the older subjects and other aged-matched controls by means of a structured interview. Blood will be collected for laboratory and genetic testing.

SUMMARY:
This study will systematically assess epigenome methylation changes in participants of the Israel multi-ethnic centenarian study cohort, which includes citizens of Israel aged 95 years and older, compared to their offspring and younger controls.

DETAILED DESCRIPTION:
The number of men and women reaching advanced age is rapidly increasing in developed countries and life expectancy has already doubled since the beginning of the last century. In parallel, the proportion of those who have survived to advanced old age without major health complications has become increasingly common. This phenomenon has led to concerted research efforts to understand the correlates and mechanisms of extended human longevity and healthy aging. For decades the public health perspective has emphasized environmental and life style factors as having beneficial effects on health and disease prevention in the general population. Important biological insights have been reached by examining the genetic basis of longevity and healthy aging, especially among individuals who demonstrate a favorable healthy aging phenotype. Epigenetics, defined as heritable changes in gene function or phenotypes, in the absence of DNA sequence changes, has revolutionized the concept of how genetics affect disease risk. Epigenetics have been shown to be associated with cancer risk and autoimmunity disorders. Moreover, epigenetic changes at specific sites appear to increase with age, hence they may serve as indices for chronological age. This background has led us to our central hypotheses that: i) epigenetic changes associated with healthy aging could serve as markers for a healthy life span, and ii) the epigenetic changes may represent one of the central mechanisms by which aging predisposes to many age-related diseases, and therefore affects healthy aging. We propose to test these hypotheses within the Israel multi-ethnic centenarian study cohort (which includes all citizens of Israel>95 years old; an estimated 1 in 5000 of the population). We will systematically assess genomic methylation changes in three major sub-groups which signifies three major points in human lifespan: Age 60±5 years (leading age of onset of age associated diseases and also considered to represent the beginning of old age, age 80±5 years (average life expectancy in the western world), and age 100±5 years (exceptional longevity). Our centenarians includes 3 subgroups: SURVIVORS: those who survive and become centenarians in spite of early onset of cognitive impairment, functional disability or major age associated diseases, such as diabetes, vascular disease or cancer, at the beginning of old age, i.e., age of 60±5 years (thus long life span but short healthy lifespan). DELAYERS: those who develop age related diseases or cognitive/physical disability much later than the control population i.e., at the age of 80±5 years instead of 60 years (therefore have a longer healthy life span). DODGERS: those who fail to develop age-related illnesses or cognitive/physical disability throughout their life span. We will compare these groups to healthy controls with no family history of longevity in two reference groups, namely 60±5 years and 80±5 years, comparing them to the survivors and delayers groups, respectively. We predict that subjects will exhibit differences in methylation at sites distinct from each other, in contrast to healthy subjects.

Accordingly our proposed goals are:

1. To characterize the Israel multi-ethnic centenarian study cohort (I-MECS).
2. To screen, catalog and annotate epigenome methylation variants in five different groups (a. Survivors, b. Delayers, c. Dodgers, d. 60±5YO healthy control, and e. 80±5YO healthy controls).
3. To validate differential methylated loci by ranking and prioritizing using Sequenom's MassARRAY.
4. Exploratory goal (depend on time and funding availability) - To establish expression patterns using a qRT-PCR (Polymerase Chain Reaction) Roche light-cycler of the candidate epigenetic loci identified in Aims 1, 2 and 3 as well as specific genes (such as deoxyribonucleic acid methyltransferase and tumor suppressor genes) in blood cells of the initially screened population.

To test our hypotheses, we propose to employ a novel high-throughput genome-wide methylation assay, namely HELPtag. Additionally, we will utilize a combination of epigenome-wide association studies (EWAS) to identify the most distinctive epigenetic loci that show greatest differential methylation. We will then perform multi-locus validation for methylation status using MassARRAY.

ELIGIBILITY:
Inclusion Criteria:

* Aged 95 years and older.
* Provide verbal consent for participation in the study.
* Cognitively able to provide consent and answer a structured questionnaire.

Exclusion Criteria:

* Not able to provide consent for participation in the study.
* Impaired consciousness.
* Unable to communicate.

Min Age: 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Subjects aged 95 years and older will form the study cohort. Control group will comprise children of the older subjects and age-matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of alleles in genes across the genome | 6 months
  Variations of frequency of alleles in study groups using dedicated software for genomic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Tzvi Dwolatzky, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, North, Israel

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared

REFERENCES:
- [Background] Brooks-Wilson AR. Genetics of healthy aging and longevity. Hum Genet. 2013 Dec;132(12):1323-38. doi: 10.1007/s00439-013-1342-z. Epub 2013 Aug 8. PMID 23925498
- [Background] Evert J, Lawler E, Bogan H, Perls T. Morbidity profiles of centenarians: survivors, delayers, and escapers. J Gerontol A Biol Sci Med Sci. 2003 Mar;58(3):232-7. doi: 10.1093/gerona/58.3.m232. PMID 12634289
- [Background] Wojdacz TK, Hansen LL. Techniques used in studies of age-related DNA methylation changes. Ann N Y Acad Sci. 2006 May;1067:479-87. doi: 10.1196/annals.1354.069. PMID 16804030